CLINICAL TRIAL: NCT06668519
Title: An Observational Study on the Clinical Application of Magnetoencephalography in Children With Neurodevelopmental Disorders
Brief Title: Magnetoencephalography in Children
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-173
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Epilepsy; Intracranial Tumors; Cerebrovascular Disease; Autism; ADHD - Attention Deficit Disorder With Hyperactivity; Neuropsychiatric Disorders; Tic Disorder, Childhood; Mental Retardation; Developmental Disabilities
Keywords: neurodevelopmental diseases; magnetoencephalography; pediatric
MeSH Terms: conditions — Epilepsy; Brain Neoplasms; Cerebrovascular Disorders; Autistic Disorder; Attention Deficit Disorder with Hyperactivity; Tic Disorders; Intellectual Disability; Developmental Disabilities | interventions — Magnetoencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with neurodevelopmental diseases
  Interventions: Other: Magnetoencephalography
- healthy children
  Interventions: Other: Magnetoencephalography

INTERVENTIONS:
Other: Magnetoencephalography — Magnetoencephalography

SUMMARY:
This study is a single-center observational clinical study, which evaluates the diagnostic value of magnetoencephalography (MEG) in the diagnosis of neurodevelopmental diseases in children, such as the localization of epileptic foci and brain functional areas, intracranial tumors, cerebrovascular diseases, autism, mental retardation, and neuropsychiatric disorders.

DETAILED DESCRIPTION:
The purpose of this study is to observe the application of magnetoencephalography (MEG) in pediatric neurodevelopmental disorders

ELIGIBILITY:
Inclusion Criteria:

1. aged 1 month-18 years old (date of investigate minus date of birth)
2. epilepsy
3. intracranial tumors
4. cerebrovascular diseases
5. autism
6. mental retardation
7. ADHD
8. tic disorder
9. neuropsychiatric disorders

Exclusion Criteria:

1.Unable to cooperate with the exam of MEG

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 1 month to 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Difference in magnetoencephalography (MEG) signal between children with neurodevelopmental diseases and healthy children | 3 years
  Acquisition of magnetoencephalography (MEG) signals based on Inclusion Criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No